CLINICAL TRIAL: NCT02725424
Title: A Randomized, Controlled Phase II Study to Compare Preoperative Chemotherapies in Locally Advanced Gastric/Gastroesophageal Cancer
Brief Title: Optimizing the Strategy for Preoperative Chemotherapy in Locally Advanced Gastric/Gastroesophageal Cancer
Acronym: MATCH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Aiping Zhou, Chief physician, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-071
Record Dates: First submitted 2016-03-11; First posted 2016-04-01 (Estimated); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — S 1 (combination); Oxaliplatin; Trastuzumab; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Her2 Positive with SOX (Active Comparator): Oxaliplatin 130 mg/m2, ivgtt, d1; S-1 twice a day depending on body surface areas (BSA) po d1-14, 80mg/day (BSA <1.25m2) ,100mg/day (BSA ≥1.25m2, <1.5 m2), 120mg/day (BSA ≥1.5m2), every 3 weeks.
  Interventions: Drug: S-1; Drug: Oxaliplatin
- Her2 Positive with SOXT (Experimental): Oxaliplatin 130 mg/m2, ivgtt, d1; S-1 twice a day depending on body surface areas (BSA) po d1-14, 80mg/day (BSA <1.25m2) ,100mg/day (BSA ≥1.25m2, <1.5 m2), 120mg/day (BSA ≥1.5m2), trastuzumab 8mg/kg (loading dose), 6mg/kg subsequently ivgtt d1, every 3 weeks.
  Interventions: Drug: S-1; Drug: Trastuzumab; Drug: Oxaliplatin
- Her2 Negative with SOX (Active Comparator): Oxaliplatin 130 mg/m2, ivgtt, d1; S-1 twice a day depending on body surface areas (BSA) po d1-14, 80mg/day (BSA <1.25m2) ,100mg/day (BSA ≥1.25m2, <1.5 m2), 120mg/day (BSA ≥1.5m2), every 3 weeks.
  Interventions: Drug: S-1; Drug: Oxaliplatin
- Her2 Negative with DOS (Experimental): Docetaxel 60 mg/m2, ivgtt, d1; Oxaliplatin 100 mg/m2, ivgtt, d1; S-1 twice a day depending on body surface areas (BSA) po d1-14, 80mg/day (BSA <1.25m2) , 100mg/day (BSA ≥1.25m2, <1.5 m2), 120mg/day (BSA ≥1.5m2), every 3 weeks.
  Interventions: Drug: S-1; Drug: Oxaliplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: S-1 — Her-2 Positive patients with SOX Oxaliplatin：130 mg/m2, iv, d1 S-1：twice a day depending on BSA po from d1-14, 80mg(BSA <1.25m2) , 100mg(BSA ≥1.25m2, <1.5 m2), 120 mg(BSA≥ 1.5m2), Every 3 weeks.
  Other Names: Oxaliplatin
Drug: Trastuzumab — Her-2 positive patients with SOXT Oxaliplatin：130 mg/m2, iv, d1 S-1：twice a day depending on BSA po from d1-14, 80mg(BSA <1.25m2) , 100mg(BSA ≥1.25m2, <1.5 m2), 120 mg(BSA≥ 1.5m2), Trastuzumab: 8mg/kg (loading dose), 6mg/kg subsequently ivgtt d1 Every 3 weeks.
  Other Names: Oxaliplatin; S-1
  Arms: Her2 Positive with SOXT
Drug: Oxaliplatin — Her-2 Positive patients with SOX Oxaliplatin：130 mg/m2, iv, d1 S-1：twice a day depending on BSA po from d1-14, 80mg(BSA <1.25m2) , 100mg(BSA ≥1.25m2, <1.5 m2), 120 mg(BSA≥ 1.5m2), Every 3 weeks.
  Other Names: S-1
Drug: Docetaxel — Her-2 Negative patients with DOS Docetaxel： 60 mg/m2, iv, d1 Oxaliplatin：100 mg/m2, iv, d1 S-1：twice a day depending on BSA po from d1-14, 80mg(BSA <1.25m2) , 100mg(BSA ≥1.25m2, <1.5 m2), 120 mg(BSA≥ 1.5m2), Every 3 weeks
  Other Names: Oxaliplatin; S-1
  Arms: Her2 Negative with DOS

SUMMARY:
This is a randomized, phase II, open-label study. The purpose of this study is to determine the optimal treatment for patients with locally advanced Gastric/Gastroesophageal Cancer according to their HER-2 expression status.

The primary endpoint of this study: major pathology response rate the second endpoints of this study: pathology complete response rate R0 resection rate Progression-free survival ( PFS) Disease -free survival (DFS) Overall survival(OS) Objective response rate(ORR) Adverse event(AE)

DETAILED DESCRIPTION:
(HER2, human epidermal growth factor receptor-2) positive patients: After 4 cycles of SOX±Trastuzumab neoadjuvant therapy, patients will continue to accept D2 surgery. The patients with R0 resection will continue to receive 4 cycles of SOX±Trastuzumab adjuvant chemotherapy. If the patients are confirmed with tumor progression before surgery, the treatment such as gastrectomy, chemoradiotherapy or second line chemotherapy should be determined by MDT team.

(HER2, human epidermal growth factor receptor-2,HER2) negative patients： After 4 cycles of DOS or SOX regimen as neoadjuvant therapy, patients will continue to accept D2 surgery. The patients with R0 resection will continue to receive then 4 cycles of DOS or SOX adjuvant chemotherapy. If the patients are confirmed with tumor progression before surgery, the treatment such as gastrectomy, chemoradiotherapy or second line chemotherapy should be determined by MDT team.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically confirmed gastric cancer or gastroesophageal junction adenocarcinoma;
2. The HER2 receptor protein status should be assessed using immunohistochemistry (IHC) and fluorescence in situ hybridization (FISH);

   * HER2 positive: IHC 3+ or IHC 2+/ FISH amplification.
   * HER2 negative: IHC 0, 1+ or IHC 2+/ FISH without amplification.
3. T3-4, any N stage, M0 of gastric or gastro-esophageal junction adenocarcinoma;
4. Chemotherapy and radiotherapy naïve.
5. Age ≥18 years;
6. ECOG(Eastern Cooperative Oncology Group ) 0-1;
7. Adequate hematological, hepatic and renal functions: absolute neutrophil count (ANC) ≥ 2.0 G/L, hemoglobin ≥ 90g/L, platelet ≥ 100 G/L; ALT and AST <1.5 times x upper limit of normal (ULN)；serum total bilirubin < 1.0 x ULN; serum creatinine < 1.0 x ULN;
8. Left ventricular ejection fraction>50%
9. Written informed consent.

Exclusion criteria:

1. Other pathology Type Other than adenocarcinoma, such as squamous cell carcinoma
2. History of allergies to drugs in the study
3. Intraperitoneal dissemination or distant metastasis
4. Digestive tract obstruction or uncontrollable recurrent bleeding ,clinical significant ascites
5. Dysphagia
6. Any cause of cirrhosis
7. Cardiac function NYHA(New York Heart Association) >I degrees
8. Previous myocardial infarction, unstable angina, stroke ,or uncontrollable Arrhythmia
9. Any surgical contraindication
10. Any chemotherapy or radiotherapy history
11. Any surgical resection history of gastric cancer
12. History of any other tumors except cured cutaneum carcinoma or carcinoma in situs of cervix
13. Any contraindication for chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
major Pathological response rate | 40 months

CONTACTS AND LOCATIONS:
Overall Officials: Ping Ai Zhou, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided